CLINICAL TRIAL: NCT00512408
Title: Long-Acting Testosterone Improves Exercise Oxygen Uptake, Insulin Resistance and Muscle Strength in Elderly Patients With Chronic Heart Failure
Brief Title: Testosterone Improves Exercise Oxygen Uptake, Insulin Resistance and Muscle Strength in Elderly Patients With Chronic Heart Failure
Status: Terminated | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Other Study IDs: 002-07
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-08

CONDITIONS: Congestive Heart Failure
Keywords: To assess the effect of a 12 week testosterone administration on maximal exercise capacity, muscle strength and insulin resistance in elderly CHF patients
MeSH Terms: conditions — Heart Failure | interventions — Testosterone

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- A
  Interventions: Drug: testosterone
- B

INTERVENTIONS:
Drug: testosterone
  Groups: A

SUMMARY:
Background: Patients with congestive heart failure (CHF) show muscle mass wasting and decreased testosterone levels. Long-term testosterone supplementation improves walking distance and glucose metabolism of patients CHF. No studies have investigated the integrated effects of testosterone on exercise oxygen uptake muscle strength and glucose metabolism in patients with CHF regardless of the presence of hypogonadism.

Aim: To assess the effect of a 12 week testosterone administration on maximal exercise capacity, muscle strength and insulin resistance in elderly CHF patients.

Methods: Seventy elderly patients with stable CHF, mean age 71 ± 8 years, ejection fraction 34 ± 1%, NYHA class II/III 38/32, were enrolled. Of these, 35 were randomized to receive testosterone therapy (through intramuscular injection every 6 week) and 35 to receive placebo both on top of maximal medical therapy. At baseline and after 12 weeks all patients underwent echocardiogram, cardiopulmonary test, 6-minute walking test (6MWT), quadriceps maximal isometric and isokinetic strength.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction (LVEF) < 40%;
* New York Heart Association (NYHA) class II or III;
* clinical stability without hospital admission for heart failure in the previous 3 months.

Exclusion Criteria:

* unstable angina or recent acute myocardial infarction,
* history of severe liver diseases
* history of severe kidney diseases
* uncontrolled hypertension
* erythrocytosis (hematocrit > 50%)
* hyperviscosity
* prostate cancer, prostate-specific antigen (PSA) greater than 3 ng/ml
* severe lower urinary tract symptoms.

Ages: 56 Years to 76 Years | Sex: Male
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: maurizio volterrani, md, Principal Investigator — IRCCS san Raffaele Cardiovascular Research Unit; giuseppe marazzi, md, Principal Investigator — IRCCS san Raffaele Cardiovascular Research Unit; massaro rosalba, md, Principal Investigator — IRCCS san Raffaele Cardiovascular Research Unit; marco miceli, Principal Investigator — IRCCS san Raffaele Cardiovascular Research Unit; caterina mammi, Principal Investigator — IRCCS san Raffaele Cardiovascular Research Unit; massimo fini, md, Principal Investigator — IRCCS san Raffaele Cardiovascular Research Unit; giuseppe rosano, md, Study Director — IRCCS san Raffaele Cardiovascular Research Unit
Locations (1):
- IRCCS San Raffaele, Rome, rome, Italy

REFERENCES:
- [Derived] Schwartz JB, Volterrani M, Caminiti G, Marazzi G, Fini M, Rosano GM, Iellamo F. Effects of testosterone on the Q-T interval in older men and older women with chronic heart failure. Int J Androl. 2011 Oct;34(5 Pt 2):e415-21. doi: 10.1111/j.1365-2605.2011.01163.x. Epub 2011 May 25. PMID 21615419